CLINICAL TRIAL: NCT02304575
Title: Quality of Life Among Testicular Cancer Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0482-14-RMC
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Testicular Neoplasms; Spermatic Cord Torsion; Varicocele; Testicular Hydrocele
MeSH Terms: conditions — Testicular Neoplasms; Spermatic Cord Torsion; Varicocele; Testicular Hydrocele | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Testicular cancer survivors: Patients treated for testicular cancer, will receive questionnaires and hormonal function measurement.
  Interventions: Other: Questionnaires; Other: Hormonal Function measurement
- Surgery for benign testicular problems: Patients treated for benign testicular conditions, will receive questionnaires and hormonal function measurement.
  Interventions: Other: Questionnaires; Other: Hormonal Function measurement
- Healthy males: Healthy volunteers, will receive questionnaires and hormonal function measurement.
  Interventions: Other: Questionnaires; Other: Hormonal Function measurement

INTERVENTIONS:
Other: Questionnaires — Questionnaires:
  For examinee: European Organization for Research and Treatment of Cancer quality of life questionnaire of 30 items and testicular cancer module of 26 items (EORTC QLQ-30 + QLQ-TC-26), Multidimensional Coping Inventory, The Meaning Test for cognitive function, cognitive orientation questionnaires.
  For partner: Multidimensional Inventory of quality of life (QoL) for Adults, Multidimensional Coping Inventory.
Other: Hormonal Function measurement — Plasma levels of: follicular stimulating hormone (FSH), luteinizing hormone (LH), thyroid-stimulating hormone (TSH), prolactin, free androgen index.

SUMMARY:
Testicular Cancer is the most prevalent malignancy among men between 20 and 34 years of age, with incidence rates rising in western countries including Israel. Cure rate of testicular cancer exceeds 90% with modern treatments. Thus issues such as quality of life (QoL), coping, effects on couple relationships, cognitive function, cognitive orientation and hormonal function become increasingly important. This study aims to assess all these issues using validated, reproducible questionnaires and hormonal plasma levels, and compare them between testicular cancer survivors and controls.

DETAILED DESCRIPTION:
The study will be conducted in RMC, Beilinson and Golda. Eligible male patient list will be drawn from the Rabin Medical Center (RMC) operation rooms' data system.

Patients will be contacted by their treating urologists over the phone or during follow-up visits and invited to take part in the research which will be conducted at RMC. The first stage of the study will include a validation of the EORTC QLQ-TC26 questionnaire in Hebrew.

Patients and partners / spouses will sign informed-consent forms and fill out questionnaires during their visit, and blood samples will be drawn on the day of questionnaire completion or no longer than 1 month from it. Spouses will be given the choice of arriving with the patient and filling-in their questionnaires at RMC, or having them mailed to their homes. Research assistants will provide assistance with the questionnaires.

Normal controls will be recruited among Tel Aviv University students, 'Achva' College students and RMS staff and asked to come to RMC for blood tests. Control subjects will be asked to answer the same cancer-related questionnaires as the patients, as fully as possible, unless the questions are irrelevant to them.

The anticipated recruitment period will be approximately 36 months. Financial incentives: a compensation of 150 NIS will be offered to healthy participants coming to RMC for blood tests under this study.

Duration of research participation: 1 or 2 encounters (the second for missing data or missing blood samples, and in the first 30 patients - for TC26 questionnaire re-validation by the EORTC requirements), during no longer than 1 month for each participant.

Measurements will be compared across the patient and 2 control groups and their correlation to hormonal function assessed.

ELIGIBILITY:
Inclusion Criteria:

Group1: Testicular cancer long-term survivors

* Male subjects between 2 to 10 years after testicular cancer diagnosis, who have completed treatment and are regarded as complete responders.
* Able to give informed consent Group 2: Benign testicular conditions patients
* Male subjects between 2 to 10 years after testicular surgery due to a benign condition.
* Able to give informed consent Group 3: Healthy Controls
* Healthy males
* Able to give informed consent Partners of males from above 3 groups
* Females or males
* In a couple relationship with a man of 1 of the above groups, for 1 year or longer.
* Able to give informed consent

Exclusion criteria:

Group1: Testicular cancer long-term survivors

* Inability to answer questionnaires (i.e due to mental impairment).
* Another malignancy, other than non-invasive skin basal cell carcinoma (BCC) or squamous cell carcinoma (SCC).
* Testicular cancer recurrence. Group 2: Benign testicular conditions patients
* Inability to answer questionnaires.
* Any history of malignancy other than non-invasive skin BCC or SCC. Group 3: Healthy Controls
* Inability to answer questionnaires.
* Any history of malignancy other than non-invasive skin BCC or SCC.
* Any history of testicular surgery or diagnosed testicular problems in adulthood or childhood.

Partners of males from above 3 groups

- Inability to answer questionnaires.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group1: Testicular cancer long-term survivors Group 2: Benign testicular conditions patients Group 3: Healthy Controls Partners of males from above 3 groups
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QLQ), as measured by the QLQ-TC26 (Testicular Cancer 26 items) questionnaire. | 2-10 years from diagnosis

SECONDARY OUTCOMES:
Hormonal function, as measured by follicular stimulating hormone (FSH) & free androgen index | 2-10 years from diagnosis
cognitive orientation score | 2-10 years from diagnosis
multidimensional coping score | 2-10 years from diagnosis
cognitive function as measured by the meaning test | 2-10 years from diagnosis
Partner's Quality of life, as measured by the multidimensional inventory of QOL for adults questionnaire | 2-10 years from diagnosis
Partner's Coping mechanism score, as measured by the Multidimensional Coping Inventory | 2-10 years from diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD PhD, Principal Investigator — Rabin MC
Locations (1):
- Rabin Medical Center, Beilinson & Hasharon Hospitals, Petah Tikva, Israel